CLINICAL TRIAL: NCT00833300
Title: Haloperidol vs Olanzapine for the Management of ICU Delirium: A Randomized Clinical Trial
Brief Title: Haloperidol vs Olanzapine for the Management of ICU Delirium
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Hall (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor-Investigator, Richard Hall, Dr. Richard Hall MD FRCPC FCCP, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDHA-RS/2009-001; Control No.:121747; File No.: 9427-C2659-22C
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Delirium; Agitation
Keywords: Delirium; Agitation; Intensive Care; Critical Care; Antipsychotics; Olanzapine; Haloperidol
MeSH Terms: conditions — Delirium; Psychomotor Agitation | interventions — Haloperidol; Olanzapine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator): Haloperidol
  Interventions: Drug: Haloperidol
- 2 (Active Comparator): Olanzapine
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Haloperidol — * 2.5 mg-10 mg IV q6h for 24 hours and 2.5 mg-5 mg IV prn, up to 40mg in 24 hours.
  * Reassess in 24 hours.
  * Delirium absent - Continue dose for 24 hours then discontinue.
  * Delirium present - Increase dose 5 mg-10 mg IV q6h for 24 hours and 2.5 mg-5 mg IV prn, up to 40 mg in 24 hours.
  * Reassess in 24 hours.
  * Delirium absent - Continue dose for 24 hours then discontinue.
  * Delirium present - Discontinue current drug therapy and select one of:
    1. Quetiapine up to 100 mg/day
    2. Risperidone up to 6 mg/day
    3. Loxapine up to 50 mg/day
    4. Methotrimeprazine up to 75 mg/day
  * Reassess in 24 hours.
  * Delirium absent - Continue for 24 hours then discontinue.
  * Delirium present - Treatment at discretion of attending physician.
  Other Names: Haldol
  Arms: 1
Drug: Olanzapine — * 2.5 mg-10 mg po/ng/og bid and 2.5 mg po/ng/og prn, up to 20 mg in 24 hours.
  * Reassess in 24 hours.
  * Delirium absent - Continue dose for 24 hours then discontinue.
  * Delirium present - Increase dose 5 mg-10 mg bid and 2.5 mg po/ng/og prn, up to 20 mg in 24 hours.
  * Reassess in 24 hours.
  * Delirium absent - Continue dose for 24 hours then discontinue.
  * Delirium present - Discontinue current drug therapy and select one of:
    1. Quetiapine up to 100 mg/day
    2. Risperidone up to 6 mg/day
    3. Loxapine up to 50 mg/day
    4. Methotrimeprazine up to 75 mg/day
  * Reassess in 24 hours.
  * Delirium absent - Continue for 24 hours then discontinue.
  * Delirium present - Treatment at discretion of attending physician.
  Other Names: Zyprexa; Zyprexa Zydis; Novo-Olanzapine; PMS-Olanzapine
  Arms: 2

SUMMARY:
The purpose of this randomized clinical trial is to determine whether haloperidol is superior to olanzapine for the treatment of ICU acquired delirium. The hypothesis is that haloperidol is in fact superior to olanzapine in treating ICU acquired delirium and sustaining delirium free time.

DETAILED DESCRIPTION:
Delirium is defined as a disturbance of consciousness characterized by an acute onset of impaired cognitive function. Although delirium is thought to be common in the Intensive Care Unit (ICU) there are few studies that have evaluated its incidences, risks and outcomes. It has been associated with increased morbidity, and mortality and increased cost to the healthcare system. In addition to the uncertainty of the incidence of ICU delirium, there is a lack of information about the effects that certain pharmacological treatments have on delirious patients.

The standard pharmacological treatments for ICU acquired delirium are haloperidol and olanzapine as they have been shown to be equivalent in reducing its incidence. However, optimal dose and regimen have not been well defined.

The rationale for this study is to determine whether haloperidol is superior to olanzapine in the treatment of ICU acquired delirium. A secondary objective is to determine the most appropriate dosing regimen for the treatmet. The role of alternative agents quetiapine, risperidone, loxapine and methotrimeprazine will also be examined in a preliminary analysis.

Patients who develop agitation or delirium as defined by an Intensive Care Delirium Checklist (ICDSC) score of greater than or equal to 4 meeting all the inclusion criteria and no exclusion criteria will be eligible for randomization. Once randomized they will be screened for ongoing agitation and delirium as well prolongation of the QTc interval greater than 440 msec, development of extrapyramidal symptoms and development of a seizure disorder.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are 18 years or older who are admitted for more than 24 hours to the ICU.
* Patients screened for delirium using the ICDSC with a score greater than or equal to 4 or with clinical manifestations of delirium.

Exclusion Criteria:

* Patients unlikely to survive 24 hours.
* Patients with a primary neurologic reason (i.e. stroke, dementia-related psychosis) for ICU admission.
* Patients with QTc interval greater than 440 msec.
* Pregnant patients.
* Patients who are breast feeding.
* Patients in whom haloperidol, or olanzapine is contraindicated.
* Patients allergic to haloperidol, olanzapine, quetiapine, risperidone, loxapine or methotrimeprazine.
* Patients who do not have a urinary catheter.
* Patients who have received haloperidol, olanzapine, quetiapine, risperidone, loxapine or methotrimeprazine within 14 days.
* Patients unable to undergo assessment (i.e. patients with developmental disability or mental incapacity prior to ICU admission).
* Prolonged (greather than 24 hours) comatose patients who have a defined structural reason for their decreased level of consciousness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Resolution of delirium as indicated by an Intensive Care Delirium Screening Checklist score of less than 4 | Every 24 hours

SECONDARY OUTCOMES:
Delirium free days (i.e. time from resolution of delirium to ICU discharge) | Every 24 hours
Incidence of treatment failure at 48 hours | 48 hours
Requirement for rescue medication | Every 24 hours
Type of rescue medication | Every 24 hours
Mortality | Time of death
If on mechanical ventilation at time delirium develops, duration of mechanical ventilation | Every 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hall, MD, FRCPC, FCCP, Principal Investigator — Nova Scotia Health Authority
Locations (2):
- Canada (2):
  - Halifax Infirmary; Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Victoria General Hospital; Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia

REFERENCES:
- [Background] Bergeron N, Skrobik Y, Dubois MJ. Delirium in critically ill patients. Crit Care. 2002 Jun;6(3):181-2. doi: 10.1186/cc1482. Epub 2002 Apr 5. PMID 12133171
- [Background] Lacasse H, Perreault MM, Williamson DR. Systematic review of antipsychotics for the treatment of hospital-associated delirium in medically or surgically ill patients. Ann Pharmacother. 2006 Nov;40(11):1966-73. doi: 10.1345/aph.1H241. Epub 2006 Oct 17. PMID 17047137
- [Background] Jaber S, Chanques G, Altairac C, Sebbane M, Vergne C, Perrigault PF, Eledjam JJ. A prospective study of agitation in a medical-surgical ICU: incidence, risk factors, and outcomes. Chest. 2005 Oct;128(4):2749-57. doi: 10.1378/chest.128.4.2749. PMID 16236951
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Pandharipande P, Shintani A, Peterson J, Pun BT, Wilkinson GR, Dittus RS, Bernard GR, Ely EW. Lorazepam is an independent risk factor for transitioning to delirium in intensive care unit patients. Anesthesiology. 2006 Jan;104(1):21-6. doi: 10.1097/00000542-200601000-00005. PMID 16394685
- [Background] Skrobik YK, Bergeron N, Dumont M, Gottfried SB. Olanzapine vs haloperidol: treating delirium in a critical care setting. Intensive Care Med. 2004 Mar;30(3):444-9. doi: 10.1007/s00134-003-2117-0. Epub 2003 Dec 19. PMID 14685663
- [Background] Plaschke K, von Haken R, Scholz M, Engelhardt R, Brobeil A, Martin E, Weigand MA. Comparison of the confusion assessment method for the intensive care unit (CAM-ICU) with the Intensive Care Delirium Screening Checklist (ICDSC) for delirium in critical care patients gives high agreement rate(s). Intensive Care Med. 2008 Mar;34(3):431-6. doi: 10.1007/s00134-007-0920-8. Epub 2007 Nov 9. PMID 17994221
- [Background] Devlin JW, Fong JJ, Schumaker G, O'Connor H, Ruthazer R, Garpestad E. Use of a validated delirium assessment tool improves the ability of physicians to identify delirium in medical intensive care unit patients. Crit Care Med. 2007 Dec;35(12):2721-4; quiz 2725. doi: 10.1097/01.ccm.0000292011.93074.82. PMID 18074477
- [Background] Rea RS, Battistone S, Fong JJ, Devlin JW. Atypical antipsychotics versus haloperidol for treatment of delirium in acutely ill patients. Pharmacotherapy. 2007 Apr;27(4):588-94. doi: 10.1592/phco.27.4.588. PMID 17381385
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Dubois MJ, Bergeron N, Dumont M, Dial S, Skrobik Y. Delirium in an intensive care unit: a study of risk factors. Intensive Care Med. 2001 Aug;27(8):1297-304. doi: 10.1007/s001340101017. PMID 11511942
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Bucerius J, Gummert JF, Borger MA, Walther T, Doll N, Falk V, Schmitt DV, Mohr FW. Predictors of delirium after cardiac surgery delirium: effect of beating-heart (off-pump) surgery. J Thorac Cardiovasc Surg. 2004 Jan;127(1):57-64. doi: 10.1016/s0022-5223(03)01281-9. PMID 14752413
- [Background] Korevaar JC, van Munster BC, de Rooij SE. Risk factors for delirium in acutely admitted elderly patients: a prospective cohort study. BMC Geriatr. 2005 Apr 13;5:6. doi: 10.1186/1471-2318-5-6. PMID 15826320
- [Background] Stein LM, Thienhaus OJ. Hearing impairment and psychosis. Int Psychogeriatr. 1993 Spring;5(1):49-56. doi: 10.1017/s1041610293001383. PMID 8499573
- [Background] Brust JC. Acute neurologic complications of drug and alcohol abuse. Neurol Clin. 1998 May;16(2):503-19. doi: 10.1016/s0733-8619(05)70074-8. PMID 9537972
- [Background] Vincent FM. The neuropsychiatric complications of corticosteroid therapy. Compr Ther. 1995 Sep;21(9):524-8. PMID 8565441